CLINICAL TRIAL: NCT06142604
Title: Single Dose Flecainide for Early Sinus Rhythm Conversion of Perioperative Atrial Fibrillation After Noncardiac Surgery (FLIP-AF): a Pilot Randomized Controlled Trial
Brief Title: Single Dose Flecainide for Early Sinus Rhythm Conversion of Perioperative Atrial Fibrillation After Noncardiac Surgery
Acronym: FLIP-AF
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Feasibility
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-FLIPAF
Record Dates: First submitted 2023-11-10; First posted 2023-11-21 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Atrial Fibrillation; Surgery
Keywords: Flecainide
MeSH Terms: conditions — Atrial Fibrillation | interventions — Flecainide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flecainide (Experimental): Participants randomized to the flecainide arm will be prescribed a single 300mg dose of oral flecainide, to be given as soon as possible after study randomization. Rate controlling drugs will be prescribed and titrated to achieve a heart rate of less than 100 beats per minute and symptom minimization.
  Interventions: Drug: Flecainide
- No flecainide (No Intervention): Participants randomized to the no flecainide arm will not be prescribed flecainide. Rate controlling drugs will be prescribed and titrated to achieve a heart rate of less than 100 beats per minute and symptom minimization.

INTERVENTIONS:
Drug: Flecainide — Single 300mg dose of oral flecainide
  Arms: Flecainide

SUMMARY:
Investigator-initiated pilot study of single dose oral flecainide versus no flecainide for the early conversion of perioperative atrial fibrillation to sinus rhythm after noncardiac surgery.

DETAILED DESCRIPTION:
FLIP-AF is a prospective, randomized, open-label trial of single dose flecainide versus no flecainide in patients with perioperative atrial fibrillation after noncardiac surgery. The primary objective is to determine whether it is feasible to conduct a large randomized controlled trial assessing the efficacy and safety of single dose flecainide in this population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Noncardiac surgery in the last 30 days requiring an overnight hospital admission;
* Presence of AF (i.e., atrial fibrillation and/or flutter) with a ventricular heart rate of ≥ 100 beats per minute at any time within 12 hours prior to randomization;
* In AF at the time of randomization; AND,
* Provided written informed consent.

Exclusion Criteria:

* History of AF without normal sinus rhythm documented within 90 days prior to randomization;
* Hemodynamic instability;
* Have any one of the following contraindications to flecainide:

  1. known left ventricular ejection fraction ≤ 40%;
  2. myocardial infarction within the last 30 days;
  3. QRS interval >140ms;
  4. allergy to flecainide;
  5. severe uncorrected hypokalemia (<2.5 mEq/L) or hyperkalemia (>6.5 mEq/L) at the time of randomization;
  6. severe acute liver dysfunction or history of advanced cirrhosis;
  7. severe renal insufficiency (eGFR ≤ 30ml/min or dialysis); OR,
  8. second or third degree atrioventricular block within the last 30 days, in the absence of a pacemaker device;
* Unable to take oral medication;
* Previously enrolled in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | through study completion, an average of six months
  Minimum recruitment rate of at least 1.5 patients per site per month
Follow-up completion rate | through study completion, an average of six months
  Completion rate of at least 90%